CLINICAL TRIAL: NCT00887861
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Two-arm Parallel-group Study of BGG492 as Monotherapy in Individuals With Refractory Partial Seizures Undergoing Inpatient Evaluation for Epilepsy Surgery
Brief Title: Efficacy of BGG492 in Individuals With Refractory Partial Seizures Undergoing Inpatient Evaluation for Epilepsy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBGG492A2202; EudraCT 2008-005065-64
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Seizures; Epilepsy
Keywords: epilepsy; seizure; monotherapy trials; partial seizure; Partial seizures and undergoing evaluation for epilepsy surgery
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGG492 (Experimental)
  Interventions: Drug: Investigational new drug, company code: BGG492
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Investigational new drug, company code: BGG492
  Arms: BGG492
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will asses the safety and efficacy of BGG492 in reducing the seizure rate in therapy-refractory partial seizures.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of partial seizures (with or without secondary generalization) and undergoing an evaluation for epilepsy surgery, based on the classification of the International League Against Epilepsy (ILAE), as modified in 1981.
2. Absence of evolving space-occupying lesions or progressive neurological diseases.
3. Have normal vital signs (systolic and diastolic blood pressure and pulse rate)
4. All female subjects must have negative pregnancy test results
5. Subjects must weigh at least 50 kg to participate in this study and must have a body mass index (BMI) within the range of 18 to 35.

Exclusion Criteria:

1. A history of frequent and/or severe status epilepticus (i.e. requiring intensive care unit treatment).
2. Current treatment with phenobarbital, primidone or zonisamide (these drugs would have to be completely washed out before study start)
3. Having discontinued chronic benzodiazepine and barbiturate therapy within 30 days prior to the study start
4. Having electrodes implanted in the brain.
5. Having evidence on physical examination, or a history of any medically significant thyroid, cardiac, respiratory, hepatic, gastrointestinal, renal, hematologic, oncologic, psychiatric or progressive neurological disorder, requiring current medical intervention/therapy likely to have a significant impact on the outcome of this study.
6. With any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs, e.g. GI surgery and/or pancreatic or liver disease
7. Having a significant illness other than epilepsy within two (2) weeks prior to initial dosing.
8. Having recent (within the last three (3) years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Measure: An efficacy of investigation drug versus Placebo in reducing the seizure rate when administered orally for up to 7days as monotherapy in patients with refractory partial seizures who are undergoing an inpatient evaluation for epilepsy | 7 days

SECONDARY OUTCOMES:
Measure:An efficacy of investing. drug vs. Pcb in reducing the seizure rate when administered orally for up to 9days (during titration monotherapy)in pts. with refractory partial seizures who are undergoing an inpatient evaluation for epilepsy surgery. | 9 days
Measure: To evaluate the safety and tolerability of investigational drug repeated dose over 9 days in patients with refractory partial seizures | 9 days
Measure: To determine the plasma levels of investigational drug in patients with refractory partial seizures. | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bielefeld
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Erlangen
  - Novartis Investigator Site, Freiburg im Breisgau
  - Novartis Investigator Site, Munich